CLINICAL TRIAL: NCT04336670
Title: Design and Implementation of a Immersive Virtual Reality Physical Exercise Program to Improve Functional Capacities in Older People.
Brief Title: Design and Implementation of a Physical Exercise Program With Virtual Reality to Improve Functional Capacities in Older People.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pablo Campo-Prieto (Other)
Collaborators: Saraiva Senior Center (Unknown)
Responsible Party: Sponsor-Investigator, Pablo Campo-Prieto, Principal Investigator, University of Vigo
Organization: University of Vigo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HEALTHYFIT-UVIGO 2020/078
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Aging; Fall; Quality of Life
Keywords: Aged; Virtual Reality Exposure Therapy; Balance; Biomedical Technology; Exercise Therapy; Physical Therapy Modalities; Quality of Life

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality group (Experimental): Immersive Virtual Reality exercise program + Usual center therapies
  Interventions: Device: Immersive Virtual Reality exercise program
- Usual activities group (Active Comparator): Usual center therapies
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Immersive Virtual Reality exercise program — Sessions with an exercise program focused in upper and low limbs movements in a virtual enviroment, all performed in standing position.
  Arms: Virtual Reality group
Other: Usual care — Usual center therapies (Physical therapy, occupational therapy..)
  Arms: Usual activities group

SUMMARY:
TITLE: Desing and implementation of a Immersive Virtual Reality exercise program to improve balance in older people

INTRO: Older people grow around the world at a faster rate than any other age group, resulting in an accelerated aging of the population and an increase in life expectancy. In response to this new reality, active aging programs and strategies are especially relevant and it based in physical activity practice, whose main objective is to maintain or improve the functionality of the person, even though the loss of balance in the elderly represents a significant difficulty in their lives, since this aspect reduces their postural control, increasing the risk of falls and injuries. Our project REVIEM (Inmersive Virtual Reality Exergaming in Olders) is a new strategy to improve the balance in older people, using a exercise program with Virtual Reality glasses for this purpose.

HYPOTHESIS: The practice of REVIEM protocol based on physical function training in older adults collaborates in the maintenance and improvement of functional capacities, reducing the number of falls and increasing their personal autonomy.

GENERAL GOALS:

1.1 Design and implement a REVIEM exercise program / protocol to improve balance in older people 1.2 Analyze the effects of this REVIEM program / protocol, in the short and medium term in institutionalized individuals.

1.3 Identify if there is a relationship between the variables that induce fragility and functional dependence and the REVIEM protocol

SPECIFIC GOALS:

2.1 Determine the REVIEM protocol to improve differential effects for 6 minutes a day (3 days a week for 10 weeks)

2.1.1 The improvement of the functional independence of individuals by improving balance, reducing the risk of falls and proper development in activities of daily living.

2.1.2 The improvement of gait. 2.1.3 The improvement of quality of life. 2.1.4 The improvement of handgrip.

2.2 Determine the parameters related to immerse virtual reality exposure. 2.2.1 Safety of the virtual reality exposure 2.2.2 Usability of the virtual reality exposure 2.2.3 Personal experiences and satisfaction of the virtual reality exposure

METHODS:

Design: Randomized controlled trial. The institutionalized elderly from the geriatric center Saraiva Senior Center in Pontevedra, Spain, will be invited to take part in the study. After they meet the selection criteria, they will be assigned to on experimental group and one control group. Information regarding sociodemographic characteristics and a clinical anamnesis of the participants will be collected.

Intervention: Two groups (experimental and control). Experimental group will perform the REVIEM protocol sessions (6 min) focused on the upper and lower limbs. (3 sessions per week for 10 weeks). All sessions will begin with a warm-up focused on the stimulation of coordination and joint mobilization, so that the body is predisposed both centrally and peripherally for the performance of the session and will end with a stretching routine accompanied by breathing cycles calm and controlled. The session will be supervised by the physiotherapist, occupational therapist or expert in physical exercise of the center.

Control group will participate in the usual activities proposed by the center management.

Assessments: 4 evaluations will be carried: initial, intermediate (at 1 month), final (at 10 weeks) and follow-up (1 month after to end the program).

The contents of the assessmentens will be:

1. Characteristics of patients: "ad hoc" record sheet that will include data on age, sex, associated pathologies and pharmacological treatment.
2. REVIEM protocol. Safety (Simulator Sickness Questionnaire), Usability (System Usability Scale) and personal experiences (Game Experience Questionnaire and "ad hoc" interview notebook)

2. Balance, gait and fall risk (Tinetti Test) 3. Functional mobility and lower limbs strength (Five times sit to stand test) 4. Functional autonomy (Timed Up and Go Test) 5. Quality of life (SF-12 Scale) 6. Handgrip (dynamometer)

Hypothesis : our findings aim to support the use of new health technologies in the field of rehabilitation and healthcare for the elderly, achieving a feasible and safety Immersive Virtual Reality exergaming program.

ELIGIBILITY:
Inclusion Criteria:

* Saraiva Senior Center members
* Signed informed consent

Exclusion Criteria:

* Comorbidity that discourages the exercise of physical exercise and that allows to carry out all the programmed evaluations.
* Mobility problems that prevent compliance with the protocol.
* Serious visual and / or auditory disturbances that impede the development of the session, as well as those with a history of vertigo, seizures or epileptic seizures to prevent exacerbations of these symptoms as potential adverse effects of Immersive Virtual Reality.
* Severe cognitive impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Simulator Sickness Questionnaire | 4 weeks
  SSQ is used for measuring users' level of sickness symptoms and is highly appreciated in VR research. Each item is rated with the scale from none, slight, moderate to severe. Through some calculations, four representative scores can be found. Nausea-related subscore (N), Oculomotorrelated subscore (O), Disorientation-related subscore (D) are the scores for the symptoms for the specific aspects. Total Score (TS) is the score representing the overall severity of cybersickness experienced by the users of virtual reality systems.
Simulator Sickness Questionnaire | 10 weeks
  SSQ is used for measuring users' level of sickness symptoms and is highly appreciated in VR research. Each item is rated with the scale from none, slight, moderate to severe. Through some calculations, four representative scores can be found. Nausea-related subscore (N), Oculomotorrelated subscore (O), Disorientation-related subscore (D) are the scores for the symptoms for the specific aspects. Total Score (TS) is the score representing the overall severity of cybersickness experienced by the users of virtual reality systems.
System Usability Scale | 4 weeks
  SUS provides a quick and reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. It allows you to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications.
System Usability Scale | 10 weeks
  SUS provides a quick and reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. It allows you to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications.
Game Experience Questionnaire (post game module) | 4 weeks
  GEQ can be applied after playing the game, several times over a longer period - also to see the changes in the experience. It is applicable for lab and field evaluation studies.Post game module - conserns experiences once a player has stopped gaming.Captures the game experience based on a number of items (such as positive affect, competence, immersion, flow, challenge).
Game Experience Questionnaire (post game module) | 10 weeks
  GEQ can be applied after playing the game, several times over a longer period - also to see the changes in the experience. It is applicable for lab and field evaluation studies.Post game module - conserns experiences once a player has stopped gaming.Captures the game experience based on a number of items (such as positive affect, competence, immersion, flow, challenge).
Tinetti Test | pre intervention
  The Tinetti Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks. Scoring of the Tinetti Assessment Tool is done on a three point ordinal scale with a range of 0 to 2. A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score, and overall balance assessment score, ad a combined gait and balance score. The maximum score for the gait component is 12 points. The maximum score for the balance component is 16 points. The maximum total score is 28 points. In general, residents who score below 19 are at a high risk for falls.
Tinetti Test | 10 weeks
  The Tinetti Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks. Scoring of the Tinetti Assessment Tool is done on a three point ordinal scale with a range of 0 to 2. A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score, and overall balance assessment score, ad a combined gait and balance score. The maximum score for the gait component is 12 points. The maximum score for the balance component is 16 points. The maximum total score is 28 points. In general, residents who score below 19 are at a high risk for falls.
Tinetti Test | 14 weeks
  The Tinetti Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks. Scoring of the Tinetti Assessment Tool is done on a three point ordinal scale with a range of 0 to 2. A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score, and overall balance assessment score, ad a combined gait and balance score. The maximum score for the gait component is 12 points. The maximum score for the balance component is 16 points. The maximum total score is 28 points. In general, residents who score below 19 are at a high risk for falls.
Five times sit to stand test | pre intervention
  FTSTS is used to objectively determine measures to provide a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements
Five times sit to stand test | 10 weeks
  FTSTS is used to objectively determine measures to provide a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements
Five times sit to stand test | 14 weeks
  FTSTS is used to objectively determine measures to provide a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements
Time Up and Go Test | pre intervention
  Standardized test to assess the basic functional mobility of elderly persons and requires both static and dynamic balance. The patient is observed and timed while he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again.
Time Up and Go Test | 10 weeks
  Standardized test to assess the basic functional mobility of elderly persons and requires both static and dynamic balance. The patient is observed and timed while he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again.
Time Up and Go Test | 12 weeks
  Standardized test to assess the basic functional mobility of elderly persons and requires both static and dynamic balance. The patient is observed and timed while he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again.
SF-12 Scale | pre intervention
  It is one of the most used questionnaires to evaluate the multidimensional health related quality of life, worldwide. The 12 items are a subset of those in the SF-36 and measures 8 concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems and mental health (psychological distress and psychological well being).
SF-12 Scale | 10 weeks
  It is one of the most used questionnaires to evaluate the multidimensional health related quality of life, worldwide. The 12 items are a subset of those in the SF-36 and measures 8 concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems and mental health (psychological distress and psychological well being).
Strengh | pre intervention
  handgrip strength
Strengh | 10 weeks
  handgrip strength
Strengh | 14 weeks
  handgrip strength

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Campo-Prieto, PT M. Sc., Principal Investigator — HealthyFit Research Group - University of Vigo
Locations (1):
- Pablo Campo-Prieto, Pontevedra, Galicia, Spain